CLINICAL TRIAL: NCT05356208
Title: Long-term Outcome After Bascom's Cleft-lift Procedure Under Tumescent Local Analgesia for Pilonidal Sinus Disease: a Cohort Study
Brief Title: Long-term Outcome After Cleft-lift for Pilonidal Sinus Disease
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSD - cleft-lift
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-04

CONDITIONS: Pilonidal Sinus
Keywords: Cleft-lift; Tumescent local analgesia
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-center cohort study of 10-year risk of treatment failure after cleft-lift under tumescent local analgesia for pilonidal sinus disease

DETAILED DESCRIPTION:
The standard treatment at Nordsjællands Hospital in Hillerød (NOH) has since 2007 been Bascom's pit-pick procedure (PP) for simple pilonidal sinus disease (PSD), while Bascom's cleft-lift procedure (CL)has been performed in complicated cases not suitable for PP operation, recurrences following previous excisions, including PP, and unhealed midline wounds.

CL has mainly been performed under tumescent local analgesia (TLA) in a day-surgery setting. TLA is well tolerated with high patient satisfaction and acceptable short-term outcomes. TLA provides a potentially higher cost-effectiveness not requiring presence of an anesthesiologist, shorter duration of the complete procedure and elimination of the risks and discomforts associated with general anesthetics.

The study is based on data of patients in a local pilonidal database. The patients in the database have all undergone surgery for pilonidal sinus disease at NOH during the period of 2007 to 2014. Data in the database has been collected prospectively up to one year following surgery and subsequently supplemented with data collected by questionnaire and telephone interviews for the period from one year follow-up and until the date of long-term follow-up. Study data were collected and managed using REDCap electronic data capture tools hosted at NOH.

Patients receive a REDCap survey per e-mail to a personal digital mailbox or are asked to participate in a telephone interview to fill out a standardized questionnaire. Patients without a personal digital mailbox receive the questionnaire by regular mail. The survey is sent out twice with a four-week interval. Only patients who do not fill out the questionnaire the first time, receive the survey a second time as a reminder. Telephone interviews are only conducted, if patients do not reply to the questionnaire received digitally or as a physical copy. The questionnaire includes questions regarding demographic characteristics, lifestyle, complications, recurrence and new interventions, pain, and cosmetic satisfaction. Medical records are reviewed to verify answers from the questionnaire if consent by the patient is given through the survey or during the telephone interview. Patients experiencing symptoms of recurrence, are offered an assessment at the hospital.

The procedure has been described previously and performed with minor modifications of the original description by John Bascom. All procedures were performed in a day-surgical setting. With the patient in the prone position, the natal cleft was opened and exposed by retraction with elastic bandage tape before the sterile surgical draping was applied. The resection area and a flap on the less affected side were outlined with the intention of 2-3 cm lateralization of the wound. A hockey incision was outlined in the distal part of the excision to achieve lateralization at the distal end of the wound. Subcutaneous TLA with a modified Klein's solution containing mepivacaine 0.8 mg/mL, adrenaline 1 µg/mL, and sodium bicarbonate 42 µg/mL in isotonic saline water was infused through a 2-inch 21-gauge needle under a pressure of approximately 300 mm hg using a pressure infusion bag. If fibrous tissue affected the subcutaneous tissue, the solution was infiltrated by a 20-ml syringe. In case of pain during surgery, a supplementary tumescent solution was administered. If acceptable analgesia could not be obtained, intravenous sedation or analgesia was administrated at the patient's request.

A flap with a thickness of approximately 7 mm was mobilized to the marked outer line to ensure tension-free tissue coverage of the excision. All primary pits in the midline were excised en-bloc, and all hair and granulation tissue in the subcutis was removed with a surgical swap or by curettage, saving as much fibrotic tissue as possible to provide padding. The retraction tape was released, and the surgical wound was closed with absorbable monofilament multilayer sutures subcutaneously with the intention of reducing any dead space in the subcutis before intracutaneous closure with polypropylene or monofilament short-term absorbable suture. A 10-French drain with no vacuum or silicon ribbon drains was placed under the flap. The wound was reinforced with strips and covered by a hydrofiber bandage. All patients received one dose of cefuroxime 1.5 g and metronidazole 1.0 g intravenously preoperatively, and cephalexin 500 mg and metronidazole 500 mg orally three times daily for three days as prophylaxis.

Risk of recurrence is analyzed using competing risk analysis as well as univariate and multivariate Cox regression analyses including the following risk factors: sex, age, smoking, BMI, relevant co-morbidities, diabetes mellitus, acne, hidradenitis, previous interventions, preoperative abscess, number of primary and secondary pits, number of lateral incisions and postoperative complications. Time to complete wound healing is analyzed by Kaplan-Meier plots. Remaining outcomes are analyzed as categorical variables using descriptive data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing pit-pick at Nordsjællands Hospital during the study period

Exclusion Criteria:

* Non-Danish residents
* Patients planned for general anesthesia were excluded

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to complex pilonidal sinus disease referred to a secondary and tertiary care hospital. Patients with history of surgery for pilonidal sinus disease are included in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure assessed by clinical assessment or by questionnaire | 10 years
  Incomplete wound healing or recurrence after complete wound healing

SECONDARY OUTCOMES:
Chronic pain related to cicatrix | 10 years
  Numerical rate scale pain score (0-10). 0 being no pain and 10 being the the worst
Cosmetic appearance of the cicatrix | 10 years
  Numerical rate scale score (1-5). 1 being worst, 5 the better

CONTACTS AND LOCATIONS:
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No
fter de-identification, individual participant data will be made available to investigators who provide a methodologically sound proposal for meta-analyses.

REFERENCES:
- [Background] Bertelsen CA. Cleft-lift operation for pilonidal sinuses under tumescent local anesthesia: a prospective cohort study of peri- and postoperative pain. Dis Colon Rectum. 2011 Jul;54(7):895-900. doi: 10.1007/DCR.0b013e31820ee852. PMID 21654258
- [Result] Svarre KJ, Serup CM, Kanstrup CTB, Kleif J, Bertelsen CA. Long-term outcome after Bascom's cleft-lift procedure under tumescent local analgesia for pilonidal sinus disease: a cohort study. Colorectal Dis. 2023 Apr;25(4):707-716. doi: 10.1111/codi.16420. Epub 2022 Nov 28. PMID 36401803